CLINICAL TRIAL: NCT00005518
Title: Epidemiology and Immunology of Hemophilia A Inhibitors
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5038; R01HL061937 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2004-08

CONDITIONS: Blood Disease; Hemophilia A
MeSH Terms: conditions — Hematologic Diseases; Hemophilia A

SUMMARY:
To determine the risk factors associated with inhibitor formation in hemophilia A and to study the mechanism of tolerance in the murine hemophilia A model.

DETAILED DESCRIPTION:
BACKGROUND:

The major hypothesis of this study is that suppression of immunoregulatory cytokines will prevent factor VIII inhibitor formation in the hemophilia A murine model: if successful, a treatment protocol could be developed for individuals identified to be at highest risk for inhibitor formation. Through this approach to the epidemiology and immunology of inhibitor formation, the health care of individuals with hemophilia may be improved.

The study is in response to a Request for Applications released in 1998 on the Immunogenetics of Inhibitor Formation in Hemophilia. .

DESIGN NARRATIVE:

A case-control study is conducted comparing prevalent hemophilia patients with inhibitors identified in the HMS Study with three age-matched controls without inhibitors to determine clinical and laboratory characteristics associated with inhibitor development. A histocompatibility study is conducted identifying patterns of HLA Class II antigens by molecular typing in hemophilic subjects identified in HMS, with and without inhibitors, which may be linked to inhibitor formation. An animal tolerance study is conducted in the hemophilia A murine model, evaluating blockade of T cell costimulatory pathways by CTLA4-Ig and anti-CD40L mAb, to prevent inhibitor formation.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-06; Study Completion 2003-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M.V. Ragni — University of Pittsburgh